CLINICAL TRIAL: NCT00886470
Title: Phase I/II Randomized Blinded Safety, Dose-determining Efficacy Trial Comparing Amnion-derived Cellular Cytokine Solution in 3 Different Regimens With Standard Care 0.9% Sodium Chloride in the Topical Treatment of Partial-thickness Burns
Brief Title: ST266 Versus Standard Care In Treating Partial Thickness Burns
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated early due to slow accrual of patients.
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACCS-PT-09.001
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Burns
Keywords: cytokines; pain; scarring; vascularity
MeSH Terms: conditions — Burns; Pain; Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ST266 1 (Experimental): Topical treatment every other day
  Interventions: Biological: ST266
- ST266 2 (Experimental): Topical treatment every 4th day
  Interventions: Biological: ST266
- ST266 3 (Experimental): Topical treatment every 7th day
  Interventions: Biological: ST266

INTERVENTIONS:
Biological: ST266 — ST266 is a clear liquid containing more than 200 proteins, cytokines, and growth factors in solution. Patients will be treated for 21 days unless both wounds have healed prior to 21 days, at which time a punch biopsy of the epithelialized area of each wound will be performed. A study evaluation visit for assessment of the biopsy site will occur on day 28 or within 7 days of the punch biopsies, whichever occurs first. Six months after the punch biopsy, the patient will return to the burn center for a final examination and photographs of the study wounds.

SUMMARY:
The objective of this protocol is to perform a safety and dose-determination efficacy clinical trial in patients having a degree of partial-thickness burn wounds. The trial will be a prospectively randomized and double-blind trial of ST266 compared with standardized care using 0.9% NaCl (normal saline) solution in the same three treatment regimens.

DETAILED DESCRIPTION:
A Phase I/II multi-center clinical trial will be performed in 99 adults with partial-thickness burns. Two similar partial-thickness burn areas in a single patient will be selected. One burn will be randomly assigned to receive either test drug ST266 or normal saline in one of three treatment regimens.

The three treatment arms will be:

1. ST266 0.01 mL/cm2 every 7th day vs. normal saline 0.01 mL/cm2 every 7th day;
2. ST266 0.01 mL/cm2 every 4th day vs. normal saline 0.01 mL/cm2 every 4th day; and
3. ST266 0.01 mL/cm2 every other day vs. normal saline 0.01 mL/cm2 every other day.

Two different preclinical studies of partial-thickness burns on guinea pigs have demonstrated accelerated epithelialization with topical treatment with ST266. Similarly, preclinical studies in Yorkshire pigs have demonstrated more rapid maturity of epithelialization and better quality healing of partial-thickness skin graft donor sites with ST266 treatment.

In the preclinical studies, ST266 given in a dose of 0.01 mL/cm2 wound area appeared to saturate the wound adequately without excess and simultaneously improve healing. In preclinical toxicity studies, the dose of 0.01 mL/cm2 was shown to be safe.

ELIGIBILITY:
Inclusion Criteria:

* A signed IRB (Institutional Review Board)- approved Informed Consent Form;
* 18 - 65 years of age;
* Two (2) similar, non-contiguous, partial-thickness burn wounds between 50 cm2 and 250 cm2 in area with blisters removed in a Total Body Surface Area(TBSA) burn of less than or equal to 40% TBSA;
* Burns must be thermal burns of flame or scald etiology;
* Patient must present to the burn center within 8 hours of injury;
* Normal creatinine and bilirubin levels;
* If capable of bearing children, patient must be using a medically accepted means of birth control and have a negative serum pregnancy test;
* Willing to participate in the clinical study and comply with the requirements of the trial.

Exclusion Criteria:

* The two (2) chosen wounds must not be full-thickness (extending through the dermis into the subcutaneous tissue);
* Thermal burn from chemical, electrical or radiation causes;
* Neither the study wound nor the comparator wound can be < 50 cm2 or >250 cm2 in size and cannot be on the face or hands;
* Patients with significant pulmonary injury, i.e., smoke inhalation injury requiring ventilator support;
* Patients with diabetes;
* Patients with any immune deficiency including current treatment with corticosteroid medication, chemotherapeutic agents, anti-viral therapy, or concurrent radiation therapy within 30 days of signing the informed consent;
* Abnormal bilirubin, liver function studies (i.e., Alanine transaminase (ALT); Aspartate transaminase (AST)> 2.0 times normal);
* Abnormal serum creatinine, receiving hemodialysis or peritoneal dialysis;
* Active cancer or a history of cancer in the 5 years prior to signing the informed consent form (history of basal cell carcinoma is allowed);
* Psychiatric condition or substance abuse which in the Investigator's opinion may pose a threat to patient compliance;
* History of non-compliance with treatment or clinical visit attendance.
* Patients whose burns were previously treated with anything other than ice, cold water or dry dressing.
* Participation in an investigational trial within 30 days of study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the percentage of each wound that has epithelialized during the 21-day treatment period comparing the ST266-treated wound with the saline-treated wound. | 21 days

SECONDARY OUTCOMES:
The number of totally epithelialized (100%) wounds in the ST266-treated wounds versus the number in the normal saline-treated wounds | 21 days
The percentage conversion to full-thickness wounds in the ST266-treated wounds versus the conversion in the normal saline-treated wounds | 21 days
Quality of healing, including pruritis, and scar hypertrophy, and reduction in pain in the ST266-treated wounds as compared to saline-treated wounds | 21 days
Quality of healing as assessed by hemoxylin and eosin staining of the punch biopsy taken on Day 21 in the ST266-treated wounds as compared to saline-treated wounds | 21 days
Assessment of change in arterial circulation using a laser Doppler from baseline to Day 21 in the ST266-treated wounds as compared to saline-treated wounds | 21 days
Determination of levels of 6 cytokines present in blood prior to treatment (baseline) and within one-hour of the first treatment for the initial 12 patients | 21 days
The primary safety endpoint will be the incidence of adverse events post-treatment. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David L Steed, MD, Study Director — Noveome Biotherapeutics, formerly Stemnion
Locations (14):
- United States (14):
  - University of South Alabama Dept. of Surgery, Mobile, Alabama
  - LAC - USC Medical Center, Los Angeles, California
  - Shands Burn Center at the University of Florida, Gainesville, Florida
  - University of South Florida / Tampa General Hospital, Tampa, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Johns Hopkins Burn Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Missouri Health Care, Columbia, Missouri
  - Acute & Critical Care Surgery Barnes Jewish Hospital, Washington University Medical Center, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - MetroHealth Medical Center, Cleveland, Ohio
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - John S. Dunn Sr. Burn Center, Houston, Texas